CLINICAL TRIAL: NCT04613310
Title: PCR and Rapid Diagnostic Test on Saliva and Nasopharyngeal Swabs for the Detection of SARS-CoV-2: a Comparative Clinical Trial
Brief Title: PCR and Rapid Diagnostic Test on Saliva and Nasopharyngeal Swabs for the Detection of SARS-CoV-2 (COVID-19)
Acronym: RaDiCo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-02269
Record Dates: First submitted 2020-10-26; First posted 2020-11-03 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: COVID-19; SARS-CoV-2; Saliva; Rapid Diagnostic Test; Antigen; PCR
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: 4 components Nasopharyngeal swab by PCR Nasopharyngeal swab by RDT Saliva by PCR Saliva by RDT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Saliva and nasopharyngeal swabs (Other): One patient will have 4 swabs taken, 2 saliva for PCR and RDT, 2 nasopharyngeal for PCR and RDT
  Interventions: Diagnostic Test: Rapid Diagnostic Test vs PCR

INTERVENTIONS:
Diagnostic Test: Rapid Diagnostic Test vs PCR — 4 swabs taken, saliva for PCR and RDT, nasopharyngeal for PCR and RDT
  Other Names: Saliva versus nasopharyngeal swab

SUMMARY:
Recent literature shows that the sensitivity of the PCR tests for the detection of SARS-CoV-2 using saliva samples is close to that using nasopharyngeal swabs. This type of sampling represents a practical advantage since it can be performed by the patient herself/himself and would thus allow to speed up the collection process. It is also less painful and could prevent the rare lesions to the nasal mucosa that can occur when using nasopharyngeal swabs.

Rapid Diagnostic Tests for the detection of SARS-CoV-2 antigens have been developed using nasophayngeal swabs and have shown very high sensitivity against PCR, ranging from 93% to 98% when based on laboratory validation, 80% when based on clinical validation.This method offers the considerable advantage to inform the patient of the test result on site, and allow the provision of appropriate recommendations on the spot of testing. The studies performed so far have been conducted using nasopharyngeal samples only. There are no data with saliva yet. It is expected that the RDT would also work on the saliva. Even if slightly less sensitive due to the fact that it detects antigens and not multiplied RNA as PCR does, RDT on saliva could better serve the public health goal to test widely and quickly and have ultimately more COVID cases detected and isolated, and hence reduced transmission.

To investigate the case detection rates of both PCR on saliva and nasopharynx and RDT on nasopharynx and saliva, the patient will be taken four samples, two swabs on saliva, one for RDT and one for PCR, and two swabs on nasopharynx, one for RDT and one for PCR. Patients who have at least one of the common symptoms and who consent to such a procedure will be recruited to compare the four results. The primary objective is to compare the case detection rates for SARS-CoV-2 of the four testing methods (two sampling types and two test types).

DETAILED DESCRIPTION:
Background:

Recent literature shows that the sensitivity of the PCR tests for the detection of SARS-CoV-2 using saliva samples is close to that using nasopharyngeal swabs. This type of sampling represents a practical advantage since it can be performed by the patient herself/himself and would thus allow to speed up the collection process. It is also less painful and could prevent the rare lesions to the nasal mucosa that can occur when using nasopharyngeal swabs.

Rapid Diagnostic Tests for the detection of SARS-CoV-2 antigens have been developed using nasophayngeal swabs and have shown very high sensitivity against PCR, ranging from 93% to 98% when based on laboratory validation, 80% when based on clinical validation.This method offers the considerable advantage to inform the patient of the test result on site, and allow the provision of appropriate recommendations on the spot of testing. The studies performed so far have been conducted using nasopharyngeal samples only. There are no data with saliva yet. It is expected that the RDT would also work on the saliva. Even if slightly less sensitive due to the fact that it detects antigens and not multiplied RNA as PCR does, RDT on saliva could better serve the public health goal to test widely and quickly and have ultimately more COVID cases detected and isolated, and hence reduced transmission.

To investigate the case detection rates of both PCR on saliva and nasopharynx and RDT on nasopharynx and saliva, patients will be taken four samples, two swabs on saliva, one for RDT and one for PCR, and two swabs on nasopharynx, one for RDT and one for PCR. Patients who have at least one of the common symptoms and who consent to such a procedure will be recruited to compare the four results. The primary objective is to compare the case detection rates for SARS-CoV-2 of the four testing methods (two sampling types and two test types).

Methods:

Procedures:

Patients fulfilling inclusion and exclusion criteria will be recruited consecutively. After confirmation of inclusion and exclusion criteria, patients will be asked whether they would be willing to provide two saliva samples and one nasopharyngeal swab in addition to that provided for routine testing. After written informed consent, patients will be asked to perform swabbing of the gingiva-buccal fold two times and a saliva sample under professional supervision, once for sending to the laboratory to perform PCR, and once for performing the RDT onsite according to manufacturer's information. They will also be taken two nasopharyngeal swabs, one for RDT and one for PCR. No coughing or sniffing prior to sample collection is required. Ideally, water should be avoided 10 minutes prior to collection. Other drinks, food, and nasal sprays should be avoided 20 minutes before sample collection.

The saliva and nasopharyngeal samples will be analysed by PCR according to the standard procedure.

The RDTs will be performed and results read according to the manufacturer information (see below). Alternatively one of the three following tests will be tested: RDT from Roche (Standard Q COVID-19, the RDT from Abbott (Panbio COVID-19 Ag) and the RDT from AAZ-LMB (COVID-VIRO).

The patient will be considered as positive for SARS-CoV-2 if any of the test results (by RDT, or PCR on saliva or nasopharynx) is positive.

ELIGIBILITY:
Inclusion Criteria:

- Outpatient aged above 18 years who reports having at least one of the following symptoms: reported cough, reported fever, reported anosmia, or reported ageusia

Exclusion Criteria:

* Unwilling or incapable of informed consent
* Hospitalized patients
* Anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 949 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of SARS-CoV-2 positive patients for the two different sampling types (saliva vs nasopharyngeal) and two methods (RDT vs PCR) . | 48 hours
  Number of SARS-CoV-2 positive patients by sampling type (saliva and nasopharyngeal swab) and analytical method (RDT and PCR)

SECONDARY OUTCOMES:
Viral loads of SARS-CoV-2 by PCR on saliva and nasopharyngeal swabs | 48 hours
  Ct values by PCR in saliva and nasopharyngeal swab

CONTACTS AND LOCATIONS:
Overall Officials: Valérie D'Acremont, MD PhD, Principal Investigator — Unisanté
Locations (1):
- Unisanté, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Schwob JM, Miauton A, Petrovic D, Perdrix J, Senn N, Gouveia A, Jaton K, Opota O, Maillard A, Minghelli G, Cornuz J, Greub G, Genton B, D'Acremont V. Antigen rapid tests, nasopharyngeal PCR and saliva PCR to detect SARS-CoV-2: A prospective comparative clinical trial. PLoS One. 2023 Feb 24;18(2):e0282150. doi: 10.1371/journal.pone.0282150. eCollection 2023. PMID 36827328